CLINICAL TRIAL: NCT06674343
Title: The Efficacy and Safety of Furmonertinib 160mg as First-line Treatment in Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) With EGFR Classical Mutations, a Prospective, Single-arm, Multicenter Clinical Study
Brief Title: Furmonertinib 160mg as First-line Treatment in Locally Advanced or Metastatic NSCLC With EGFR Classical Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-24PJ1180
Record Dates: First submitted 2024-07-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-07

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: advanced or metastatic non-small cell lung cancer; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): Furmonertinib 160mg, once daily, orally
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 160mg, once daily, orally. Other Names: AST2818

SUMMARY:
To evaluate the efficacy, safety, recurrence site, recurrence pattern and resistance mechanism of 160mg furmonertinib as first-line therapy in advanced or metastatic non-small cell lung cancer (NSCLC) patients with EGFR classical mutations(19Del or L858R).

DETAILED DESCRIPTION:
To evaluate the PFS, ORR, DCR, OS, CNS ORR CNS DCR, CNS PFS, safety, recurrence site, recurrence pattern and resistance mechanism of 160mg furmonertinib as first-line therapy in advanced or metastatic non-small cell lung cancer (NSCLC) patients with EGFR classical mutations(19Del or L858R).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, Male or Female
* Histologically or cytologically confirmed locally advanced or metastatic lung adenocarcinoma not amenable to curative surgery or radiotherapy;
* Patients have been confirmed by local laboratory to have one of the following EGFR mutations: 19Del or L858R (single or compound)
* Patients had locally advanced NSCLC or metastatic NSCLC without any systemic antitumor therapy
* Having at least one measurable lesion (in accordance with RECIST1.1). Note: measurable lesion can neither be subject to local therapy as radiotherapy nor used for biopsy in screening period; if there is only one measurable lesion, this lesion will be permitted to be biopsied. However, the baseline radiological examination can be performed for this lesion at least 14 days after biopsy
* Adequate organ function as shown in the laboratory test, including: (1) ANC >= 1.5 x 10^9/L; PLT >= 100 x 10^9/L; HGB >= 90 g/L; (2) TBIL <= 1.5 times ULN, AST and ALT <= 2.5 times ULN (with liver metastasis, TBIL <= 3 times ULN, AST and ALT <= 5 times ULN); (3) CrCL >= 50 mL/min (according to Cockcroft-Gault formula);
* ECOG PS 0-1, and there was no obvious disease deterioration within 2 weeks prior to screening
* Life expectancy > 12 weeks after the first dose of investigational product
* Female of childbearing age are not pregnant and have no pregnancy plan. Female subjects at childbearing age and male subjects agree to take effective contraceptive measures during the study and within 6 months after drug discontinuation
* Being able to understand and voluntarily participate in the study, and sign the informed consent form.

Exclusion Criteria:

* NSCLC with predominant squamous cell histology, small cell lung cancer or neuroendocrine carcinoma indicated by histology or cytology test
* Patients with other driver oncogenes (ALK fusion, ROS1 fusion, RET rearrangement, BRAF mutation, NTRK fusion, MET mutation, KRAS mutation, but not TP53, RB1, BRAC mutation, etc.);
* Expected to receive other anti-tumor therapy other than the investigational product during the study
* Having received the following therapies: (1) Having been irradiated for > 30% bone marrow or a large area within 4 weeks prior to the first dose of investigational product; (2) Having received major surgery within 4 weeks prior to the first dose of investigational product or plan to receive major surgery during the study with exception of the surgical procedures to establish vascular access, biopsy through mediastinoscopy or thoracoscopy; (3) Use of a potent CYP3A4 inhibitor within 7 days prior to the first dose of investigational product or a potent CYP3A4 inducer within 21 days prior to the first dose of investigational product; use of the traditional Chinese medicine or traditional Chinese medicine preparation with tumor indication, or traditional Chinese medicine or traditional Chinese medicine preparation with adjuvant anti-tumor effect within two weeks prior to the first dose of investigational product or expected to be required during the study; (4) Having participated in the clinical trial and received the investigational product or device within 4 weeks or at least 5 half-lives prior to the first dose of investigational product; (5) Having received other anti-tumor drugs within 14 days prior to the first dose of investigational product;
* Concurrent spinal cord compression or symptomatic brain metastasis
* The toxicity caused by previous anti-tumor therapy has not recovered to <= CTCAE grade 1 (CTCAE 5.0) (except alopecia, sequelae of previous platinum-related neurotoxicity) or the level specified in the inclusion/exclusion criteria;
* Unstable pleural effusion or peritoneal effusion with obvious symptoms; those with stable clinical symptoms for at least 14 days after drainage of pleural effusion or ascites will be eligible
* Having a history of other malignant tumor, or other concurrent malignant tumors (except those that have undergone radical operation and have no recurrence within 5 years post operation, e.g. cervical carcinoma in situ, basal cell carcinoma of skin and papillary thyroid carcinoma)
* Previous interstitial lung disease (ILD), drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy; or having the clinical manifestations of suspected interstitial lung disease
* Having severe or uncontrolled systemic disease requiring treatment that is considered by investigators as ineligible for the study, including hypertension, diabetes, chronic heart failure (NYHA Functional Classification III-IV), unstable angina pectoris, myocardial infarction within one year, active hemorrhagic disease, etc.
* QTc > 470 ms on ECG at resting state
* Clinically significant prolonged QT interval or other arrhythmia or clinical status considered by investigators that may increase the risk of prolonged QT interval; for example, complete left bundle branch block, degree III atrioventricular block, congenital long QT syndrome, serious hypokalemia, or current use of drugs that may lead to prolonged QT interval
* Serious gastrointestinal dysfunction, or disease that may affect the intake, transportation or absorption of investigational product
* Infectious disease requiring intravenous medication
* Known history of mental disease or drug abuse, and currently having an attack or still taking drugs
* Known or suspected allergy to Furmonertinib or other components of its preparation
* Female subjects or female partners of male subjects who are pregnant or lactating, or plan to be pregnant during the study
* Poor compliance, inability to comply with the study procedures, restriction or requirements
* Other conditions that are considered by investigators as unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Freae Survival (PFS) | Approximately 24 months after the first patient begin study treatment
  The time from the first dose of the study drugs to the progression of the disease or death for any reason according to RECIST 1.1 by investigator

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 weeks after the last patient begin study treatment
  Rate of subjects whose tumors are assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.
Disease Control Rate (DCR) | Approximately 12 weeks after the last patient begin study treatment
  Rate of subjects whose tumors are assessed as CR, PR or stable disease (SD) according to RECIST 1.1
Overall survival (OS) | Approximately 24 months after the last patient begin study treatment
  The time from the first dose of the study drugs to the death for any reason according to RECIST 1.1
Central Nervous System Objective Response Rate (CNS ORR) | Approximately 12 weeks after the last patient begin study treatment
  Rate of subjects whose CNS tumors are assessed as complete response(CR) or partial response(PR) according to RECIST 1.1
Central Nervous System Disease Control Rate (CNS DCR) | Approximately 12 weeks after the last patient begin study treatment
  Rate of subjects whose CNS tumors are assessed as CR, PR or stable disease (SD) according to RECIST 1.1
Central Nervous System Progression Free Survival (CNS PFS) | Approximately 24 months after the first patient begin study treatment
  The time from the first dose of the study drugs to the progression of the CNS disease or death for any reason according to RECIST 1.1
Adverse Events (AEs) | From the start of study drug to 28 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided